CLINICAL TRIAL: NCT04299724
Title: Safety and Immunity Evaluation of A Covid-19 Coronavirus Artificial Antigen Presenting Cell Vaccine
Brief Title: Safety and Immunity of Covid-19 aAPC Vaccine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Collaborators: Shenzhen Third People's Hospital (Other); Shenzhen Second People's Hospital (Other)
Responsible Party: Principal Investigator, Lung-Ji Chang, President, Shenzhen Geno-Immune Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-20002
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Treat and Prevent Covid-19 Infection
Keywords: Lentiviral vector, Covid-19/aAPC vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Injection of Covid-19/aAPC vaccine (Experimental)
  Interventions: Biological: Pathogen-specific aAPC

INTERVENTIONS:
Biological: Pathogen-specific aAPC — The subjects will receive three injections of 5x10^6 each Covid-19/aAPC vaccine via subcutaneous injections.

SUMMARY:
In December 2019, viral pneumonia (Covid-19) caused by a novel beta-coronavirus (SARS-CoV-2) broke out in Wuhan, China. Some patients rapidly progressed and suffered severe acute respiratory failure and died, making it imperative to develop a safe and effective vaccine to treat and prevent severe Covid-19 pneumonia. Based on detailed analysis of the viral genome and search for potential immunogenic targets, a synthetic minigene has been engineered based on conserved domains of the viral structural proteins and a polyprotein protease. The infection of Covid-19 is mediated through binding of the Spike protein to the ACEII receptor, and the viral replication depends on molecular mechanisms of all of these viral proteins. This trial proposes to develop universal vaccine and test innovative Covid-19 minigenes engineered based on multiple viral genes, using an efficient lentiviral vector system (NHP/TYF) to express viral proteins and immune modulatory genes to modify artificial antigen presenting cells (aAPC) and to activate T cells. In this study, the safety and immune reactivity of this aAPC vaccine will be investigated.

DETAILED DESCRIPTION:
Background:

The 2019 discovered new coronavirus, SARS-CoV-2, is an enveloped positive strand single strand RNA virus. The number of SARS-CoV-2 infected people has increased rapidly and WHO has warned that the pandemic spread of Covid-19 is imminent and would have disastrous outcomes. Covid-19 could pose a serious threat to human health and the global economy. There is no vaccine available or clinically approved antiviral therapy as yet. This study aims to evaluate the safety and immune reactivity of a genetically modified aAPC universal vaccine to treat and prevent Covid-19.

Objective:

Primary study objectives: Injection of Covid-19/aAPC vaccine to volunteers to evaluate the safety.

Secondary study objectives: To evaluate the anti- Covid-19 reactivity of the Covid-19/aAPC vaccine.

Design:

1. Based on the genomic sequence of the new coronavirus SARS-CoV-2, select conserved and critical structural and protease protein domains to engineer lentiviral minigenes to express SARS-CoV-2 antigens.
2. The Covid-19/aAPC vaccine is prepared by applying lentivirus modification including immune modulatory genes and the viral minigenes, to the artificial antigen presenting cells (aAPCs). The Covid-19/aAPCs are then inactivated for proliferation and extensively safety tested.
3. The subjects receive a total of 5x10^ 6 cells each time by subcutaneous injection at 0, 14 and 28 days. The subjects are followed-up with peripheral blood tests at 0, 14, 21, 28 and 60 days until the end of the test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and Covid-19-positive volunteers
* The interval between the onset of symptoms and randomized is within 7 days in Covid-19 patients. The onset of symptoms is mainly based on fever. If there is no fever, cough or other related symptoms can be used;
* White blood cells ≥ 3,500/μl, lymphocytes ≥ 750/μl;
* Human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV) or tuberculosis (TB) test negative;
* Sign the Informed Consent voluntarily;

Exclusion Criteria:

* Subject with active HCV, HBV or HIV infection.
* Subject is albumin-intolerant.
* Subject with life expectancy less than 4 weeks.
* Subject participated in other investigational vaccine therapies within the past 60 days.
* Subject with positive pregnancy test result.
* Researchers consider unsuitable.

Ages: 6 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-15 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of vaccine events | Measured from Day 0 through Day 28
  Frequency of vaccine events such as fever, rash, and abnormal heart function.
Frequency of serious vaccine events | Measured from Day 0 through Day 28
  Frequency of serious vaccine events
Proportion of subjects with positive T cell response | 14 and 28 days after randomization

SECONDARY OUTCOMES:
28-day mortality | Measured from Day 0 through Day 28
  Number of deaths during study follow-up
Duration of mechanical ventilation if applicable | Measured from Day 0 through Day 28
  Duration of mechanical ventilation use in days. Multiple mechanical ventilation durations are summed up
Proportion of patients in each category of the 7-point scale | 7,14 and 28 days after randomization
  Proportion of patients in each category of the 7-point scale, the 7-category ordinal scale that ranges from 1 (discharged with normal activity) to 7 (death)
Proportion of patients with normalized inflammation factors | 7 and 14 days after randomization
  Proportion of patients with different inflammation factors in normalization range
Clinical improvement based on the 7-point scale if applicable | 28 days after randomization
  A decline of 2 points on the 7-point scale from admission means better outcome. The 7-category ordinal scale that ranges from 1 (discharged with normal activity) to 7 (death)
Lower Murray lung injury score if applicable | 7 days after randomization
  Murray lung injury score decrease more than one point means better outcome. The Murray scoring system range from 0 to 4 according to the severity of the condition

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, Principal Investigator — Shenzhen Geno-Immune Medical Institute
Locations (1):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No